CLINICAL TRIAL: NCT03208088
Title: Clinical Evaluation of Multifocal Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5935
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (10):
- Sequence 1 (Experimental): etafilcon A Test Lens 1 (experimental) / etafilcon A Test Lens 2 (experimental) / etafilcon A Test Lens 3 (experimental) / etafilcon A Control Lens (Active Comparator) / etafilcon A Test Lens 4 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 2 (Experimental): etafilcon A Test Lens 2 (experimental) / etafilcon A Test Lens 3 (experimental) / etafilcon A Test Lens 1 (experimental) / etafilcon A Test Lens 4 (experimental) / etafilcon A Control Lens (Active Comparator)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 3 (Experimental): etafilcon A Test Lens 3 (experimental) / etafilcon A Test Lens 4 (experimental) / etafilcon A Test Lens 2 (experimental) / etafilcon A Control Lens (Active Comparator) / etafilcon A Test Lens 1 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 4 (Experimental): etafilcon A Test Lens 4 (experimental) / etafilcon A Control Lens (Active Comparator) / etafilcon A Test Lens 3 (experimental) / etafilcon A Test Lens 2 (experimental) / etafilcon A Test Lens 1 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 5 (Experimental): etafilcon A Control Lens (Active Comparator) / etafilcon A Test Lens 1 (experimental) / etafilcon A Test Lens 4 (experimental) / etafilcon A Test Lens 2 (experimental) / etafilcon A Test Lens 3 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 6 (Experimental): etafilcon A Test Lens 4 (experimental) / etafilcon A Test Lens 3 (experimental) / etafilcon A Control Lens (Active Comparator) / etafilcon A Test Lens 2 (experimental / etafilcon A Test Lens 1 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 7 (Experimental): etafilcon A Control Lens (Active Comparator) / etafilcon A Test Lens 4 (experimental) / etafilcon A Test Lens 1 (experimental) / etafilcon A Test Lens 3 (experimental) / etafilcon A Test Lens 2 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 8 (Experimental): etafilcon A Test Lens 1 (experimental) / etafilcon A Control Lens (Active Comparator) / etafilcon A Test Lens 2 (experimental) / etafilcon A Test Lens 4 (experimental / etafilcon A Test Lens 3 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 9 (Experimental): etafilcon A Test Lens 2 (experimental) / etafilcon A Test Lens 1 (experimental) / etafilcon A Test Lens 3 (experimental / etafilcon A Control Lens (Active Comparator) /etafilcon A Test Lens 4 (experimental)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens
- Sequence 10 (Experimental): etafilcon A Test Lens 3 (experimental) / etafilcon A Test Lens 2 (experimental) / etafilcon A Test Lens 4 (experimental) / etafilcon A Test Lens 1 (experimental / etafilcon A Control Lens (Active Comparator)
  Interventions: Device: etafilcon A Investigational Toric Multifocal Contact Lens

INTERVENTIONS:
Device: etafilcon A Investigational Toric Multifocal Contact Lens — Test Lens 1
Device: etafilcon A Investigational Toric Multifocal Contact Lens — Test Lens 2
Device: etafilcon A Investigational Toric Multifocal Contact Lens — Tes Lens 3
Device: etafilcon A Investigational Toric Multifocal Contact Lens — Test Lens 4
Device: etafilcon A Investigational Toric Multifocal Contact Lens — Control Lens

SUMMARY:
This is a double-masked, bilateral, randomized, non-dispensing clinical trial. The study lenses will be worn in a bilateral and random fashion using a 5x5 crossover Williams design with 5 lens types and 5 periods. The subjects will wear each pair of lenses for approximately 15 minutes with a 15 minute wash-out between each pair. Two lens types will be fit at the first visit and three lens types will be fit at the second visit. Using a computer-generated randomization scheme, each subject will randomly be assigned to 1 of 10 unique sequences of the 5 lens types. Randomization will be stratified by site.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol
  3. The subject must be between 40 and 70 years of age.
  4. The subject's distance refraction must be in the range of -1.50 D to -4.50 D.
  5. The subject's refractive cylinder must be -1.00 to -1.50 D in each eye
  6. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye
  7. The subject must have best corrected visual acuity of 20/20-3 or better in each eye
  8. Subjects must own a wearable pair of spectacles if required for their distance vision
  9. The subject must be an adapted soft contact lens wearer in both eyes (ie, worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month or more duration)
  10. The subject must already be wearing a presbyopic contact lens correction (eg, reading spectacles over contact lenses, multifocal or monovision contact lenses, etc) or if not respond positively to at least one symptom on the "Presbyopic Systems Questionnaire".

Exclusion Criteria:

1. Ocular or systemic allergies or disease, or use of medication which might interfere with contact lens wear
2. Pregnancy or lactation
3. Currently diagnosed with diabetes
4. Infectious diseases (eg, hepatitis, tuberculosis) or an immune-suppressive disease (eg, HIV).
5. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear
6. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions
7. Any previous, or planned, ocular or intraocular surgery (eg, radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc)
8. A history of amblyopia, strabismus or binocular vision abnormality
9. Any ocular infection or inflammation
10. Any ocular abnormality that may interfere with contact lens wear
11. Use of any ocular medication, with the exception of rewetting drops
12. History of herpetic keratitis
13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment
14. Employee of clinical site (eg, Investigator, Coordinator, Technician).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Golden Optometric Group, Whittier, California
  - Bay Hill Eye Care, Orlando, Florida
  - Lee & Leong Doctors of Optometry, Kahului, Hawaii
  - Spectrum Eyecare, Jamestown, New York
  - Sacco Eye Group, Vestal, New York
  - Miamisburg Vision Care, Miamisburg, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 96 subjects were enrolled in this study, of which 91 subjects were assigned at least 1 study lens, 5 subjects failed to meet all eligibility criteria. Of the total assigned subjects, 88 completed the study, while 3 were discontinued.
Pre-assignment Details: Subjects were randomized to 1 of 10 unique lens sequences.
Groups:
- Test 3/Test 2/Test 4/Test 1/Control: Subjects randomized to this sequence received the following treatments in order: Test 3 in period 1, Test 2 in period 2, Test 4 in period 3, Test 1 in period 4, Control in period 5.
- Test 3/Test 4/Test 2/Control/Test 1: Subjects randomized to this sequence received the following treatments in order: Test 3 in period 1, Test 4 in period 2, Test 2 in period 3, Control in period 4, Test 1 in period 5.
- Test 1/Control/Test 2/Test 4/Test 3: Subjects randomized to this sequence received the following treatments in order: Test 1 in period 1, Control in period 2, Test 2 in period 3, Test 4 in period 4, Test 3 in period 5.
- Test 1/Test 2/Control/Test 3/Test 4: Subjects randomized to this sequence received the following treatments in order: Test 1 in period 1, Test 2 in period 2, Control in period 3, Test 3 in period 4, Test 4 in period 5.
- Control/Test 1/Test 4/Test 2/Test 3: Subjects randomized to this sequence received the following treatments in order: Control in period 1, Test 1 in period 2, Test 4 in period 3, Test 2 in period 4, Test 3 in period 5.
- Control/Test 4/Test 1/Test 3/Test 2: Subjects randomized to this sequence received the following treatments in order: Control in period 1, Test 4 in period 2, Test 1 in period 3, Test 3 in period 4, Test 2 in period 5.
- Test 2/Test 3/Test 1/Test 4 /Control: Subjects randomized to this sequence received the following treatments in order: Test 2 in period 1, Test 3 in period 2, Test 1 in period 3, Test 4 in period 4, Control in period 5.
- Test 2/Test 1/Test 3/Control/Test 4: Subjects randomized to this sequence received the following treatments in order: Test 2 in period 1, Test 1 in period 2, Test 3 in period 3, Control in period 4, Test 4 in period 5.
- Test 4/Test 3/Control/Test 2/Test 1: Subjects randomized to this sequence received the following treatments in order: Test 4 in period 1, Test 3 in period 2, Control in period 3, Test 2 in period 4, Test 1 in period 5.
- Test 4/Control/Test 3/Test 1/Test 2: Subjects randomized to this sequence received the following treatments in order: Test 4 in period 1, Control in period 2, Test 3 in period 3, Test 1 in period 4, Test 2 in period 5.
Period: Period 1
Arm/Group | Test 3/Test 2/Test 4/Test 1/Control | Test 3/Test 4/Test 2/Control/Test 1 | Test 1/Control/Test 2/Test 4/Test 3 | Test 1/Test 2/Control/Test 3/Test 4 | Control/Test 1/Test 4/Test 2/Test 3 | Control/Test 4/Test 1/Test 3/Test 2 | Test 2/Test 3/Test 1/Test 4 /Control | Test 2/Test 1/Test 3/Control/Test 4 | Test 4/Test 3/Control/Test 2/Test 1 | Test 4/Control/Test 3/Test 1/Test 2
Started | 10 | 9 | 10 | 9 | 9 | 9 | 8 | 10 | 8 | 9
Completed | 10 | 9 | 10 | 9 | 9 | 9 | 8 | 10 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Test 3/Test 2/Test 4/Test 1/Control | Test 3/Test 4/Test 2/Control/Test 1 | Test 1/Control/Test 2/Test 4/Test 3 | Test 1/Test 2/Control/Test 3/Test 4 | Control/Test 1/Test 4/Test 2/Test 3 | Control/Test 4/Test 1/Test 3/Test 2 | Test 2/Test 3/Test 1/Test 4 /Control | Test 2/Test 1/Test 3/Control/Test 4 | Test 4/Test 3/Control/Test 2/Test 1 | Test 4/Control/Test 3/Test 1/Test 2
Started | 10 | 9 | 10 | 9 | 9 | 9 | 8 | 10 | 8 | 9
Completed | 10 | 9 | 10 | 9 | 9 | 9 | 8 | 10 | 7 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Test 3/Test 2/Test 4/Test 1/Control | Test 3/Test 4/Test 2/Control/Test 1 | Test 1/Control/Test 2/Test 4/Test 3 | Test 1/Test 2/Control/Test 3/Test 4 | Control/Test 1/Test 4/Test 2/Test 3 | Control/Test 4/Test 1/Test 3/Test 2 | Test 2/Test 3/Test 1/Test 4 /Control | Test 2/Test 1/Test 3/Control/Test 4 | Test 4/Test 3/Control/Test 2/Test 1 | Test 4/Control/Test 3/Test 1/Test 2
Started | 10 | 9 | 10 | 9 | 9 | 9 | 8 | 10 | 7 | 9
Completed | 10 | 9 | 10 | 8 | 9 | 9 | 8 | 10 | 7 | 9
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Test Article | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Test 3/Test 2/Test 4/Test 1/Control | Test 3/Test 4/Test 2/Control/Test 1 | Test 1/Control/Test 2/Test 4/Test 3 | Test 1/Test 2/Control/Test 3/Test 4 | Control/Test 1/Test 4/Test 2/Test 3 | Control/Test 4/Test 1/Test 3/Test 2 | Test 2/Test 3/Test 1/Test 4 /Control | Test 2/Test 1/Test 3/Control/Test 4 | Test 4/Test 3/Control/Test 2/Test 1 | Test 4/Control/Test 3/Test 1/Test 2
Started | 10 | 9 | 10 | 8 | 9 | 9 | 8 | 10 | 7 | 9
Completed | 10 | 9 | 10 | 7 | 9 | 9 | 8 | 10 | 7 | 9
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Test Article | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Test 3/Test 2/Test 4/Test 1/Control | Test 3/Test 4/Test 2/Control/Test 1 | Test 1/Control/Test 2/Test 4/Test 3 | Test 1/Test 2/Control/Test 3/Test 4 | Control/Test 1/Test 4/Test 2/Test 3 | Control/Test 4/Test 1/Test 3/Test 2 | Test 2/Test 3/Test 1/Test 4 /Control | Test 2/Test 1/Test 3/Control/Test 4 | Test 4/Test 3/Control/Test 2/Test 1 | Test 4/Control/Test 3/Test 1/Test 2
Started | 10 | 9 | 10 | 7 | 9 | 9 | 8 | 10 | 7 | 9
Completed | 10 | 9 | 10 | 7 | 9 | 9 | 8 | 10 | 7 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who were administered study article and completed all required study visits.
Groups:
- Completed Subjects: All subjects who were administered study article and completed all required study visits.
Arm/Group | Completed Subjects
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 26
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 7
  Black or African American | 7
  White | 73
  Other | 1
Region of Enrollment [Number; unit: Participants]
  United States | 88

OUTCOME MEASURES:

1. Primary Outcome: Overall Handling Comparison Between Test 1/Test 2 and Control
Description: Overall handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 15 minutes
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test 1: Subjects that wore the Test 1 lens in either the first, second, third, fourth, or fifth period of the study.
- Test 2: Subjects that wore the Test 2 lens in either the first, second, third, fourth, or fifth period of the study.
- Control: Subjects that wore the Control lens in either the first, second, third, fourth, or fifth period of the study.
Arm/Group | Test 1 | Test 2 | Control
Number analyzed (Participants) | 67 | 67 | 67
units on a scale | 57.1 (21.34) | 53.3 (22.47) | 52.3 (23.88)
Statistical Analysis 1: Comparison: Test 1 vs Control; Test type: Non-Inferiority — The non-inferiority of the Test lens relative to the Control will be concluded if the lower confidence limit of LSM difference is above the non-inferiority margin -5; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = 5.9, 95% CI 2-sided [0.1 to 11.6], Standard Error of Mean 2.92 — LS Mean difference was calculated as Test 1 - Control
Statistical Analysis 2: Comparison: Test 2 vs Control; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = 2.1, 95% CI 2-sided [-4.0 to 8.1], Standard Error of Mean 3.06 — LS Mean difference was calculated as Test 2 - Control

2. Secondary Outcome: Overall Handling Comparison Between Test 3/Test 4 and Control
Description: as for outcome 1
Time Frame: 15 minutes
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test 3: Subjects that wore the Test 3 lens in either the first, second, third, fourth, or fifth period of the study.
- Test 4: Subjects that wore the Test 4 lens in either the first, second, third, fourth, or fifth period of the study.
Arm/Group | Test 3 | Test 4 | Control
Number analyzed (Participants) | 67 | 67 | 67
units on a scale | 50.7 (22.59) | 49.1 (22.83) | 52.3 (23.88)
Statistical Analysis 1: Comparison: Test 3 vs Control; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean difference = -1.5, 95% CI 2-sided [-7.5 to 4.6], Standard Error of Mean 3.06 — LS Mean difference was calculated as Test 3 - Control
Statistical Analysis 2: Comparison: Test 4 vs Control; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean = -3.4, 95% CI 2-sided [-9.0 to 2.3], Standard Error of Mean 2.88 — LS Mean difference was calculated as Test 4 - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 week per subject.
Arm/Group | Test 1 | Test 2 | Test 3 | Test 4 | Control
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90 | 0/90 | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/90 | 0/89 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/90 | 0/89 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT03208088/Prot_SAP_000.pdf